CLINICAL TRIAL: NCT01518569
Title: Effect of Ulinastatin on Postoperative Systemic Inflammatory Response in Cardiac Surgery
Brief Title: Ulinastatin's Anti-inflammatory Reaction in Cardiac Surgery
Acronym: ulistin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KUH1160040
Record Dates: First submitted 2012-01-20; First posted 2012-01-26 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Cardiovascular Disease
Keywords: ulinastatin; systemic inflammation; cardiac surgery; cardiopulmonary bypass
MeSH Terms: conditions — Cardiovascular Diseases | interventions — urinastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): normal saline, same amount, iv
  Interventions: Drug: placebo
- ulinastatin (Active Comparator): 5000 unit/kg iv
  Interventions: Drug: ulinastatin

INTERVENTIONS:
Drug: ulinastatin — ulinastatin 5000 unit/kg iv before the initiation of CPB
  Other Names: ulistin
  Arms: ulinastatin
Drug: placebo — placebo (the same amount of normal saline) iv before the initiation of CPB
  Other Names: normall saline
  Arms: placebo

SUMMARY:
The purpose of the present study is to determine whether ulinastatin, urinary anti-trypsin inhibitor, attenuates cardiopulmonary bypass (CPB)-activated systemic inflammatory response in cardiac surgery with CPB.

Serial measurements and analysis of several inflammatory cytokines (bactericidal permeability increasing protein, interleukin-6, tumor necrosis factor-α)as well as markers of cardiac injury, renal impairment and oxygenation profile will be performed to determine ulinastatin's efficacy.

DETAILED DESCRIPTION:
Applying aortic cross-clamp (ACC) and cardiopulmonary bypass (CPB) for cardiac surgery produces variable systemic inflammatory reactions. As a common complication of those reactions, pulmonary dysfunction, which usually indicated by postoperative hypoxemia, is frequently associated with cardiac surgery employing CPB and has been used as a major predictor of morbidity and mortality.

Circulating humoral and cellular factors are involved in the development of the systemic inflammatory reactions including organ dysfunction. So far, many studies analyzed the concentration of inflammatory marker (cytokine) to determine the degree of systemic inflammatory responses in various conditions.

Ulinastatin has anti-inflammatory activity and suppresses the infiltration of neutrophils. Previous studies suggested ulinastatin's cytoprotective effect against ischemia-reperfusion injury in major organs and its inhibition of inflammatory marker production.

The purpose of the present study is to determine ulinastatin's possible protective efficacy of in attenuating CPB-activated systemic inflammatory response regarding postoperative cardiac, renal and pulmonary dysfunction in cardiac surgery with CPB. Serial measurements and analysis of several inflammatory cytokines, such as bactericidal permeability increasing protein (BPI), interleukin (IL)-6, tumor necrosis factor (TNF)-α, as well as markers of cardiac injury, renal impairment and oxygenation profile, such as creatine kinase-MB (CK-MB), troponin I (TnI), C-reactive protein (CRP), arterial O2 tension /inspired O2 fraction (PaO2/FiO2 ratio), will be performed to this purpose.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac surgery employing CPB

Exclusion Criteria:

* urgent/emergency surgery,
* previous heart surgery,
* combined CABG and valve surgery,
* age > 75 yrs,
* left ventricular ejection fraction < 0.45,
* diabetes treated with insulin,
* active gastropathic disorder,
* treatment for chronic obstructive pulmonary disease,
* preoperative use of steroids
* postoperative re-operation due to bleeding control
* pre and postoperative renal replacement therapy
* left ventricular assist device implantation

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
bactericidal permeability increasing protein | 5-30 min before the end of anesthesia
interleukin-6 | 5-30 min before the end of anesthesia
tumor necrosis factorTNF-α | 5-30 min before the end of anesthesia

SECONDARY OUTCOMES:
Creatine kinase-MB | before anesthesia, 24 hour after the end of anesthesia
troponin I | before anesthesia, 24 hour after the end of anesthesia
C-reactive protein | before anesthesia, 24 hour after the end of anesthesia
serum creatinine | before anesthesia, 24 hour after the end of anesthesia
PaO2/FiO2 ratio | before anesthesia, 24 hour after the end of anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Nakanishi K, Takeda S, Sakamoto A, Kitamura A. Effects of ulinastatin treatment on the cardiopulmonary bypass-induced hemodynamic instability and pulmonary dysfunction. Crit Care Med. 2006 May;34(5):1351-7. doi: 10.1097/01.CCM.0000215110.55899.AE. PMID 16540949
- [Background] Hill GE. Cardiopulmonary bypass-induced inflammation: is it important? J Cardiothorac Vasc Anesth. 1998 Apr;12(2 Suppl 1):21-5. PMID 9583572